CLINICAL TRIAL: NCT03578211
Title: Impact of Decision Aids on Bariatric Surgery Choice: A Randomized Controlled Trial
Brief Title: Impact of Decision Aids on Bariatric Surgery Choice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, SU YEN-HAO, Director of Metabolic and Weight Management Center, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: N201804032
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DAs group (Experimental): Shared decision making using decision aids
  Interventions: Behavioral: Shared decision making with decision aids
- Control group (No Intervention): Standard oral explanation guided with booklets

INTERVENTIONS:
Behavioral: Shared decision making with decision aids — For obese patients, we use shared decision making with decision aids to help them choose the suitable types of bariatric surgery.
  Arms: DAs group

SUMMARY:
Sleeve gastrectomy, Roux-en-Y gastric bypass, laparoscopic gastric banding, and bioenteric intragastric balloon insertion are common types of bariatric surgeries. These treatment strategies have diverted outcomes in body weight loss, metabolic diseases control, surgical complications, and life quality improvement. Thus, shared decision making (SDM) is necessary to aid patients to choose an appropriate treatment that suits thier needs. Investigators have developed a decision aids (DAs) and plan to conduct a randomized controlled trial (RCT) to evaluate its impact on obese patients. The measurements include a battery of interview-based questionnaires and evaluations of decision regret and knowledge improvement. Investigators expect the DAs would benefit the intervention group in the aspects of knowledge, communication and anxiety status during and after their treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) ≧ 32 kg / m2 with obesity-related comorbidity
2. Body mass index (BMI) ≧ 37 kg / m2

Exclusion Criteria:

1. Endocrine system abnormalities in patients
2. Drug abuse or mental illness
3. Major organ dysfunction and can accept surgery
4. Patients cannot understand Chinese
5. Age less than 20 years old or more than 70 years old

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-05-16 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
Decisional conflict | One week after intervention
  Total scores of decisional conflict scale

SECONDARY OUTCOMES:
Decision regret | 3 month after bariatric surgery
  Total scores of decision regret

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Hao Su, MD, Principal Investigator — Metabolic and Weight Management Center, Shuang-Ho Hospital
Locations (1):
- Taipei Medical University-Shuang Ho Hospital, New Taipei City, Zhonghe District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes